CLINICAL TRIAL: NCT03964168
Title: An Outcomes Study to Determine the Reasons Patients on Biologic Therapy Discontinue Treatment and Fail to Follow-up With Their Providers
Status: Completed | Type: Observational
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PTC05
Record Dates: First submitted 2019-05-14; First posted 2019-05-28 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Biological Factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biologic Therapy: Patient's who received and discontinued a biologic therapy
  Interventions: Drug: Biologic Agent

INTERVENTIONS:
Drug: Biologic Agent — Patients who discontinued a bioloic agent

SUMMARY:
Patient interviews to evaluate the reason patients discontinue biologic therapy and/or fail to follow up with provider.

DETAILED DESCRIPTION:
Retrospective chart review and patient interviews to evaluate the reason patients discontinue biologic therapy and/or fail to follow up with provider. This research intends to improve the continuity of care by determining why patients stop therapy and what can be done to improve their experience with the provider, pharmaceutical companies and specialty pharmacies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years of age.
* Was receiving first or second biologic therapy
* Has not had a follow up with treating physician in ≥ 9 months

Exclusion Criteria:

* Actively receiving biologic therapy

  * Was not receiving first or second biologic therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female adults ≥ 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Determine the most common reason for discontinuation | 5 years
  Tally number of patients who discontinued due to adverse events, insurance issues or category other.

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No